CLINICAL TRIAL: NCT05153135
Title: Description of Treatment Patterns and Description and Comparison of Healthcare Resource Utilization and Costs of Women With Metastatic HR+/HER2- Breast Cancer Treated With CDK4/6 Inhibitors
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLEE011AUS65
Record Dates: First submitted 2021-11-29; First posted 2021-12-10 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Metastatic Breast Cancer
Keywords: Metastatic breast cancer,; CDK4/6,; health resource utilization,; healthcare costs,; treatment patterns
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; palbociclib; abemaciclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Ribociclib: Participants who initiated CDK4/6i therapy
  Interventions: Drug: Ribociclib
- Palbociclib: Participants who initiated CDK4/6i therapy
  Interventions: Drug: Palbociclib
- Abemaciclib: Participants who initiated CDK4/6i therapy
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Ribociclib — Participants who initiated CDK4/6i therapy
  Groups: Ribociclib
Drug: Palbociclib — Participants who initiated CDK4/6i therapy
  Groups: Palbociclib
Drug: Abemaciclib — Participants who initiated CDK4/6i therapy
  Groups: Abemaciclib

SUMMARY:
The study was an observational, retrospective cohort design, using US administrative insurance claims data, to better understand Healthcare resource utilization (HRU) and healthcare costs among women with mBC initiated on a CDK4/6 inhibitor.

DETAILED DESCRIPTION:
This study used an observational, retrospective cohort design, using US administrative insurance claims data, previously employed in an existing project, to better understand HRU and healthcare costs among women with mBC initiated on a CDK4/6 inhibitor.

Adult women with HR+/HER2- mBC initiated on a CDK4/6 inhibitor were included in the study and were stratified into cohorts based on the first CDK4/6 inhibitor they received (i.e., abemaciclib, palbociclib, or ribociclib), regardless of the line of therapy and menopausal status.

The initiation of the first CDK4/6 inhibitor was defined as the index date. The index treatment was defined as the CDK4/6 inhibitor initiated on the index date (i.e., abemaciclib, palbociclib, or ribociclib).

The 6-month period preceding the index date was considered as the baseline period, and was used to measure patient characteristics.

Outcomes were measured between the index date and 1) the end of the study period (persistence, switch, HRU, costs) OR 2) the end of the index treatment (adherence, dose modification, frequency of monitoring), as relevant. The end of the study period was defined as the earliest occurrence between the end of continuous enrollment and the end of data availability.

ELIGIBILITY:
Inclusion Criteria:

- Evidence of treatment with a CDK4/6 inhibitor regardless of the line of therapy.

The initiation of the first CDK4/6 inhibitor was defined as the index date, and the first CDK4/6 inhibitor initiated was defined as the index treatment

* BC diagnosis: Two diagnosis codes of BC (International Classification of Diseases, 9th Revision, Clinical Modification [ICD-9-CM]: 174.xx and International Classification of Diseases, 10th Revision, Clinical Modification [ICD-10-CM]: C50.xx [excluding C50.x2 - male BC]) on two medical service claims separated by at least 30 days
* Metastatic disease diagnosis: At least two medical claims for a secondary neoplasm (ICD-9-CM codes: 196.xx-197.xx, 198.xx, ICD-10-CM codes: C77.xx, C78.xx, C79.xx) on separate dates, with the first one occurring no more than 30 days before the first diagnosis for BC
* HR+/HER2-: At least one prescription fill or administration of an ET (anastrazole, exemestane, ethinyl estradiol, fulvestrant, fluoxymesterone, letrozole, megestrol acetate, tamoxifen, or toremifene), HR+/HER2- therapy (everolimus), or CDK4/6 inhibitor (i.e., abemaciclib, palbociclib, or ribociclib) at any time following the diagnosis of BC, and no claims for treatments indicated for HER2+ BC, including trastuzumab, lapatinib, afatinib, pertuzumab, or ado-trastuzumab, at any time in the data period
* Women of at least 18 years of age as of the index date
* At least 6 months of continuous health plan coverage prior to and at least 1 month of continuous health plan coverage after the index date

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study analyses were conducted among HR+/HER2- women with at least one claim for treatment with CDK4/6 inhibitor for mBC
Study Population: Study analyses were conducted among HR+/HER2- women with at least one claim for treatment with CDK4/6 inhibitor for mBC
Sampling Method: Non-Probability Sample
Enrollment: 4320 (Actual)
Dates: Start 2020-05-08 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Number of inpatient (IP) admissions | From the index date defined as initiation of CDK4/6 inhibitor to the end of follow-up i.e. approximately 6 months (Q1/2001 - Q3/2018)
  Healthcare Resource Utilization (HRU) was measured between index date and end of follow-up, and was separately measured during the studied line of therapy, and after the studied line of therapy. Because women have different durations of follow-up, the number of events were reported as the average total number of visits per patient-per-6-months (PPP6M). HRU PPP6M was defined as the total number of visits or services for a patient occurring during the relevant period, reported on a six-month basis.
Number of IP days | From the index date defined as initiation of CDK4/6 inhibitor to the end of follow-up i.e. approximately 6 months (Q1/2001 - Q3/2018)
  HRU was measured between index date and end of follow-up, and was separately measured during the studied line of therapy, and after the studied line of therapy. Because women have different durations of follow-up, the number of events were reported as the average total number of visits per patient-per-6-months (PPP6M). HRU PPP6M was defined as the total number of visits or services for a patient occurring during the relevant period, reported on a six-month basis.
Number of days with durable medical equipment (DME) services | From the index date defined as initiation of CDK4/6 inhibitor to the end of follow-up i.e. approximately 6 months (Q1/2001 - Q3/2018)
  HRU was measured between index date and end of follow-up, and was separately measured during the studied line of therapy, and after the studied line of therapy. Because women have different durations of follow-up, the number of events were reported as the average total number of visits per patient-per-6-months (PPP6M). HRU PPP6M was defined as the total number of visits or services for a patient occurring during the relevant period, reported on a six-month basis.
Number of days with emergency department (ED) visits | From the index date defined as initiation of CDK4/6 inhibitor to the end of follow-up i.e. approximately 6 months (Q1/2001 - Q3/2018)
  HRU was measured between index date and end of follow-up, and was separately measured during the studied line of therapy, and after the studied line of therapy. Because women have different durations of follow-up, the number of events were reported as the average total number of visits per patient-per-6-months (PPP6M). HRU PPP6M was defined as the total number of visits or services for a patient occurring during the relevant period, reported on a six-month basis.
Number of days with outpatient (OP) services or visits | From the index date defined as initiation of CDK4/6 inhibitor to the end of follow-up i.e. approximately 6 months (Q1/2001 - Q3/2018)
  OP services included:
  * Home care services
  * Skilled nursing facility services
  * Office visits
  * Ambulatory surgical center visits
  * Other OP services
Other medical services | From the index date defined as initiation of CDK4/6 inhibitor to the end of follow-up i.e. approximately 6 months (Q1/2001 - Q3/2018)
  In addition to the all-cause HRU components, specific condition-related HRU was also analyzed. Conditions considered included those frequently encountered in clinical trials of CDK4/6 inhibitors. This included the number of days with medical services, number of IP days, number of non-IP days, and proportion of women with at least one medical service associated with a diagnosis for the following conditions:
  * Thrombolic events (e.g., thrombophlebitis/deep vein thrombosis)
  * Pulmonary embolism
  * QT prolongation events
  * Infections
  * Anemia
  * Neutropenia
  * Leukopenia
  * Thrombocytopenia
Total healthcare costs (medical service + pharmacy costs) | From the index date defined as initiation of CDK4/6 inhibitor to the end of follow-up i.e. approximately 6 months (Q1/2001 - Q3/2018)
  Medical service costs included:
  IP costs, ER costs, OP costs, DME costs, Laboratory test costs, Medical drug administration costs and OP costs - excluding drug administration costs
  Pharmacy costs (pharmacy costs covered by pharmacy benefits) included:
  CDK4/6 inhibitor costs, Endocrine and chemotherapy costs and Other drug costs

SECONDARY OUTCOMES:
Treatment patterns | From the index date defined as initiation of CDK4/6 inhibitor to the end of follow-up i.e. approximately 6 months (Q1/2001 - Q3/2018)
  Treatment patterns included:
  * Treatment persistence
  * Treatment switches
  * Treatment adherence (proportion of days covered, while on treatment)
  * Dose modification (dose decrease, dose increase)
  * Use of concomitant medication
Monitoring | From the index date defined as initiation of CDK4/6 inhibitor to the end of follow-up i.e. approximately 6 months (Q1/2001 - Q3/2018)
  electrocardiogram [EKG], hematologic tests, hepatic function tests, imaging

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

REFERENCES:
- See also: Results for CLEE011AUS65 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17887